CLINICAL TRIAL: NCT01312597
Title: Effects of Flavonoids on Cognitive Performance in Healthy Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Biochemistry, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UReading-2011-01
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Neurodegeneration
Keywords: Flavonoid; Cognitive performance; Cognitive function; Executive function; fMRI; Cerebral blood flow; Acute
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fruit beverage (Experimental)
  Interventions: Other: Fruit juice beverage
- Control beverage (Experimental)
  Interventions: Other: Fruit juice beverage

INTERVENTIONS:
Other: Fruit juice beverage — 500ml fruit juice beverage, single dose per visit
  Other Names: Tropicana Ruby Breakfast; Copella English Apple; Robinson's Lemon Barley Water

SUMMARY:
The purpose of this study is to investigate changes in cerebral blood flow, blood flavonoid levels, brain-derived neurotrophic factor, vascular reactivity and cognitive performance in young adults as a result of acute administration of a fruit-derived flavonoid-rich or flavonoid-poor drink.

DETAILED DESCRIPTION:
There has recently been an increasing interest in the potential of flavonoids, plant derived compounds found in foods such as fruit and vegetables, to ameliorate age-related cognitive decline. Research suggests that flavonoids improve memory and learning, possibly as a result of their anti-oxidant, anti-inflammatory and neuroprotective effects for example by increasing cerebral blood flow, protecting vulnerable neurons, enhancing existing neuronal function or by stimulating neuronal function. The research will initially involve a randomised cross-over human dietary intervention trial using two flavonoid-rich drinks (flavanone-rich and flavanone-poor) to investigate changes in cerebral blood flow in young adults (n=6; age range 18-30 years). Changes in cognitive performance and measures of serum BDNF levels will then be investigated in a second randomised cross-over trial using the intervention drink showing the greatest effect on cerebral blood flow in young adults (n=24; age range 18-30 years) and using a range of sensitive tests of executive function. The study is designed to measure acute effects of types of flavonoid supplementation and, as well as the primary cognitive outcome, will assess flavonoid/metabolite and BDNF (brain-derived neurotrophic factor) levels in blood and changes in vascular reactivity.

ELIGIBILITY:
Inclusion Criteria:

* MMSE between 26 and 30
* 18-30 years of age
* Native or good English speaker
* Normal BMI/body fat composition
* No significant vision, hearing or language problems
* Able to consume the beverages

Exclusion Criteria:

* Any form of disease/major mental illness/chronic fatigue syndrome
* On medication for hypertension/elevated lipids/diabetes
* On medication known to impact endothelial function
* Gall bladder/gastrointestinal abnormalities
* Sensitivity to orange or apple
* High consumer of fruit, vegetables, fruit beverages
* High consumer of caffeine or alcohol
* Consumer of illegal substances
* Vegetarian/vegan/other dieter/vigorous exerciser
* Use of antibiotics in the previous 8 weeks
* Consumer of dietary supplements

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Executive function | change in attention between baseline and 2h
  45-minute computer-based test battery of executive function tasks administered twice per visit day, at 0 hours (baseline) and 2 hours post-intervention. Visit days are at least one week apart.

SECONDARY OUTCOMES:
Cerebral blood flow | change in attention between baseline and 2h
  Non-invasive fMRI (arterial spin labelling) is conducted pre- and post-intervention at 3 time-points: 0 (baseline), and 2 and 5 hours post-intervention on 3 study days at least one week apart

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom